CLINICAL TRIAL: NCT03560284
Title: Marathon and Half Marathon Runners, Older Than 70 Years Old: Who Are They?
Acronym: MAHMROT70YO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7054
Record Dates: First submitted 2018-06-13; First posted 2018-06-18 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Follow-up Care
Keywords: Marathon; Half Marathon; Runners; Ederly; Aging process; Sport Addiction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Through this study, the investigators intend to describe the profile of marathon and half marathon runners older than 70 years old, in terms of medical, social and psychological characteristics.

First, in order to acquire a better knowledge of these aged runners: who they are; on a medical, social and psychological point of view; to figure out their motivations; to assess the impact on their life, their health and aging process.

Then, in order to be able to offer them a better medical care, in terms of prevention, treatment and follow-up care.

ELIGIBILITY:
Inclusion Criteria:

* Older than 70 years old
* Marathon or Half marathon runner
* To give an agreement to use medical datas for research study

Exclusion Criteria:

- Refusal to give an agreement to participate

Min Age: 70 Years | Sex: All
Age Groups: Older Adult
Study Population: Marathon and half marathon runners older than 70 years old
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of medical, social and psychological characteristics via a questionnare | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service Geriatrie - Soins de Suite Et Readaptation, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No